CLINICAL TRIAL: NCT04138069
Title: Effects of Imposed Pursed Lips Breathing on Breathing Pattern, Dyspnea and Pulmonary Function Test at Rest and During Exercise in COPD Patients
Brief Title: Imposed Pursed Lip Breathing at Rest and During Exercise In COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00228 Madeeha Shafeeq
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: COPD
Keywords: COPD; Pursed Lips Breathing; Dyspnea; Pulmonary Function Test (PFT); Aerobic Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLB+Aerobic Bicycling (Experimental): Pursed Lip Breathing + Aerobic Bicycling
  Interventions: Other: PLB+Aerobic Bicycling
- Aerobic Bicycling (Active Comparator): Only Aerobic bicycling
  Interventions: Other: Aerobic Bicycling

INTERVENTIONS:
Other: PLB+Aerobic Bicycling — Combination of Breathing control and Purse lips breathing technique for 5 minutes at the start of session.
  Purse lips breathing with aerobic bicycling for 8 minutes
  Arms: PLB+Aerobic Bicycling
Other: Aerobic Bicycling — Breathing control for 5 minutes at the start of session.
  Aerobic bicycling for 8 minutes
  Arms: Aerobic Bicycling

SUMMARY:
A randomized control trial was conducted at physiotherapy department of Pakistan Railway General Hospital from July 2017 to Dec 2017. 30 patients with stable COPD were enrolled in the study on the basis of inclusion and exclusion criteria. The participants were randomly assigned into two groups, Group A= interventional group, Group B = control group through toss and coin method using non-probability convenient sampling technique and written consent was obtained from each patient participated in the study. From 30 patients 15 patients were randomly allocated to each group, Group A: Interventional (n= 15), Group B: Control (n=15). 1 patient in control group B was dropout because he didn't come for follow up. Overall 29 patients were evaluated for study as in Group A, interventional (n=15) and Group B control (n=14).Patients in group A were performed breathing control at the start of session and then Purse lips breathing technique during aerobic bicycling for 8 min while in group B patients first perform breathing control and then aerobic bicycling for 8 min. Subjects in both experimental and control group underwent spirometry and baseline vitals, such as Respiratory rate, blood pressure, and oxygen saturation, at rest and at the completion of session was noted. Borg scale of dyspnea also used to rate the level of dyspnea at rest and at the end of session. Clinical COPD Questionnaire (CCQ) was used at 1st and final week of evaluation. It was 6 weeks training protocol, with three days per week session was given to the patient.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a main and growing worldwide prevailing disease that has lacking consideration from medical practitioners. COPD is self-imposed by cigarette smoking and underlying pathology is commonly irreparable. This is main reason of morbidity and mortality in under developing countries, so quick response is necessary to be aware of disease signs and symptoms to provide valuable impediment and management programs.

In U.S public survey the way prevalence of COPD has figure out by questioning adult population in case they had one of seventeen pulmonary diseases in previous months. Asthma, bronchitis and emphysema listed in these 17 diseases to approximate the cases for prevalence of disease. In era of 2000, approx. 10 million people diagnosed with COPD by doctor. Along this calculation large ratio of COPD-ers left over under diagnosed. In different countries the occurrence rate varies from 3.5% in Hong Kong and Singapore to 6.7% in Vietnam. Taken as a whole the prevalence rate is higher in Asian Pacific countries about 6.3% as compared to World Health Organisation (WHO) report data that hypothesized the figure of 3.8%.

Dyspnea is a main cause for seek medical advice or referral to pharmacotherapy and pulmonary rehabilitation regimes to lessen the inflammation and spasm of airways in addition to self management approach for example breathing retraining techniques. COPD patients have inadequate exhalation time because of increased resistance in the airways with increase chance of collapse. While doing exercise airflow limitation exacerbates that leads to air trapping with shortened exhalation phase. This is noticeable by increase in expiratory lung volumes which causes reduction in exercise capacity that might be restricted by fatigue of their lower limb muscles other than the ventilatory causes. The disease severity can be decided through the intenseness of breathlessness therefore the primary aim of COPD management is dyspnea reduction.

Commonly used strategy for ventilatory pattern training is purse lips breathing technique (PLB). PLB is supposed to alter the ventilatory pattern as a result of that breathlessness is decreased. The action of PLB technique is to improve exhalation and prevent airway obstruction. The patient performs expiration actively by means of partly opened mouth by applying pressure of 5cm of water (H2O).

PLB reduces rapid and prolong breathing and causes increased level of Carbon dioxide (CO2) in alveoli. These improved levels may dilate the airway smooth muscles and V/Q ratio and O2 in circulation. PLB is worked by generating back pressure in airways in a way to open up the narrowed airways. It is also create positive pressure during expiratory phase to prolong the exhalation time in order to decrease expiratory lung volumes and increase in tidal volume.

Patients with emphysema and bronchial atelectasis tried to perform PLB the expired air volume increased as compared to forced exhalation. This proposed that patient expires in a relaxed manner with PLB which causes less air trapping and also reduced dynamic hyperinflation.

In 2012 a randomized control study conducted on 14 stable COPD patients to rule out the effects of imposed purse lips breathing on exercise tolerance. In this study it has been shown that at rest PLB improves gaseous exchange, breathing pattern and lessen the respiratory rate near to normal.As in COPD patients' diaphragm hyperinflate due to air trapping by performing this breathing technique, diaphragm brings to a vantage point.

In COPD metabolic disruption in skeletal muscles is a main factor for exercise intolerance. Previous Investigators compared the upper and lower limb activities in COPD patients presented with obvious dyspnea and limited active daily living (ADLs). In COPD-ers due to decreased strength and endurance are correlated with early sarcopenia, reduced capacity of aerobic exercises and rapid collection of lactic acid while doing exercise these factors possible culprits for muscle fatigue. Aerobic training is well known and consistent in the improvement of disease symptoms, exercise tolerance and quality of life in patients with COPD. According to data of various studies cycle ergometer (CET) is commonly used training to increase strength and endurance in lower limb musculature. In one study results CET can cause physiological effects on COPD patients thought to improve O2 uptake & minute tidal volume with reduction in pulse rate, sensation of breathlessness and muscle fatigue.

In Pakistan about 6-7 million people have suffering due to COPD and death rate is 71 for each 10000 population. Although the demand for such strategies is considerable but at the same time the facility to grant these services is deprived. When talk about data on application of purse lips breathing technique in COPD patients, very few researches are found in Pakistan. Currently in Peshawar work on chest physiotherapy for worsening symptoms of COPD is reported. If the implication of these techniques in symptoms free period of disease this might be cause improvement in health related quality of life. The present study is to determine the effects of imposed purse lips breathing technique on dyspnea, breathing pattern and pulmonary function testing during rest and exercise in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* COPD stage 2 and 3 patients [based on "Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria]

Exclusion Criteria:

* neurological disorder and
* cardiovascular disorder
* Impaired lower limbs mobility

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-25 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 6th week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 6th week
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters.
Peak Expiratory Flow (PEF) | 6th week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.

SECONDARY OUTCOMES:
Breathing Pattern | 6th weeks
  Changes from the baseline, Breathing pattern was measured through observation and countercheck with respiratory rate which was taken by researcher by observing chest movements counting the breaths for one minute.

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MsCPPT, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No